CLINICAL TRIAL: NCT04080622
Title: A Randomized Trial to Evaluate the Efficacy of Selenium for the Prevention of Chemotherapy-induced Mucositis During Autologous Stem Cell Transplantation.
Brief Title: Evaluate the Efficacy of Selenium for the Prevention of Chemotherapy-induced Mucositis During Autologous Stem Cell Transplantation.
Acronym: AutoSelenium
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018-005033-21
Record Dates: First submitted 2019-09-02; First posted 2019-09-06 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Mucositis Oral; Stem Cell Transplant Complications
MeSH Terms: conditions — Stomatitis | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Usual care
  Interventions: Drug: Placebos
- Selenium (Active Comparator): Usual care + selenium 300 µg/day (IV infusion)
  Interventions: Drug: Selenium

INTERVENTIONS:
Drug: Selenium — Selenium 300 µg/day (IV infusion)
  Arms: Selenium
Drug: Placebos — NaCl 0,9% (IV infusion)
  Arms: Placebo

SUMMARY:
Chemotherapy-induced mucositis is an important complication after autologous stem cell transplantation. It is mainly responsible for pain and dysphagia requiring opioids and artificial nutrition. It can also induce infectious complications. A few medication has demonstrated efficacy in this setting. It has been suggested that selenium can reduce the intensity of mucositis due to its antioxydant activity. The investigators therefore perform a randomized study to confirm this preliminary data.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients receiving autologous stem cell transplantation for lymphoma or myeloma.
* Signed informed consent.

Exclusion Criteria:

* Autologous stem cell transplantation for another medical condition than lymphoma or myéloma.
* Intolerance to selenium.
* High selenium levels before study.
* Pregnancy or patients breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2023-10-08 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of severe oral mucositis (grade 3-4) | 31 months

SECONDARY OUTCOMES:
Incidence of any grade oral mucositis | 31 months
Number of days with severe oral mucositis | 31 months
Incidence of infectious complications | 31 months
Number of days with artifical nutrition | 31 months
Number of days with opioids | 31 months
Duration of hospitalization | 31 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, Maine et Loire, France

IPD SHARING:
Plan to Share IPD: Undecided